CLINICAL TRIAL: NCT01238510
Title: Comparison Between Provisional Versus Routine Kissing Balloon Technique After Main Vessel Crossover Stenting for Bifurcated Lesions.
Acronym: PROTECT-SB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Saiseikai Yokohama City Eastern Hospital (Other)
Responsible Party: Principal Investigator, Masahiro Yamawaki, Cardiology, Saiseikai Yokohama City Eastern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009009
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- Provisional fKBT (Active Comparator): Stent technique that final kissing balloon technique(fKBT) is performed if side branch flow was aggravated to TIMI0-2 after stent deployment
  Interventions: Procedure: stent technique: Provisional fKBT
- Routine fKBT (Active Comparator): Stent technique that fKBT was mandatory irrespective of side branch flow after stenting.
  Interventions: Procedure: stent technique: Routine fKBT

INTERVENTIONS:
Procedure: stent technique: Provisional fKBT — Provisional use of fKBT only when SB flow is aggravated to TIMI0-2 after stenting for non-left main bifurcation.
  Additional stenting for SB is recommended if residual stenosis (>50% in visual) or TIMI flow grade (<TIMI 3) was seen at SB after fKBT.
  Stent type: Everolimus-eluting stent only
  Arms: Provisional fKBT
Procedure: stent technique: Routine fKBT — Mandatory use of fKBT irrespective of SB flow after stenting for non-left main bifurcation. Additional stenting for SB is recommended if residual stenosis (>50% in visual) or TIMI flow grade (<TIMI 3) was seen at SB after fKBT.
  Stent type: Everolimus-eluting stent only
  Arms: Routine fKBT

SUMMARY:
In the setting of single stent strategy for treatment of bifurcation, we investigate to compare simple strategy as "provisional final kissing balloon technique(fKBT)" to complex one as "routine FKBT", focusing on actual myocardial ischemia assessed by scintigraphy in 7-month and to examine optimal endpoint of side branch ostium.

DETAILED DESCRIPTION:
Final kissing balloon technique (FKBT) is effective and accepted technique for the treatment of bifurcation. However, in complex lesion or anatomy, much procedure-time and contrast media are needed to accomplish this technique. Recent FFR study for jailed side branch (SB) demonstrated that angiographic severe stenosis at SB ostium includes "pseudo-stenosis" and stent-deployment jailing SB without FKBT has comparable impact on clinical outcome with FKBT strategy. Considering simple technique for bifurcation, we sought to investigate to compare "provisional FKBT" with "routine FKBT", focusing on actual myocardial ischemia assessed by scintigraphy in 7 month and to examine optimal endpoint of SB ostium.

ELIGIBILITY:
Inclusion Criteria:

(Patient) Patient who has angina or documented ischemia, Patients who are eligible for drug eluting stent, Age >=18, Patient who received informed consent, Patient who can receive dipyridamole-stress-technetium scintigraphy.

(Lesion) Non-left main bifurcation except for Medina class (0,0,1), De-Novo lesion, Vessel diameter in visual (main vessel>2.5mm, side branch >2.0mm), SB lesion length <5mm in visual estimate, MB lesion length < 46mm in visual, TIMI 3 in main vessel as well as side branch,

Exclusion Criteria:

(Patient) Patients who is pregnant, Patient contraindicated for antiplatelet therapy, Patients whose ejection fraction is less than 30%, Patients who has renal dysfunction, creatinine >=2.3, Patients who has live dysfunction, Patients who cannot agree with informed consent, Patient whose life expectancy is less than 1 year, Patients contraindicated for dipyridamole-stress-technetium scintigraphy.

(Lesion) Target site of acute myocardial infarction, Left main disease, In-Stent restenosis lesion, Bypass graft, Chronic total occlusion, Main vessel reference diameter >4.5mm, Bifurcation lesion that needs intended 2 stent strategy, Highly tortus and calcified lesion,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Rate of positive dipyridamole stress technetium scintigraphy | 7 month

SECONDARY OUTCOMES:
Composite of major cardiac adverse events(MACE) | 8 month
  Including cardiac death,myocardial infarction, stent thrombosis and target vessel revascularization
Angiographic restenosis rate in main vessel | 8 month
Fluoroscopic time | after procedure
Amount of contrast media | after procedure
Number of stent and wire use | after procedure
Diameter stenosis and late loss in side branch | 8 month
Regional summed difference score | 7 month

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Yamawaki, MD,PhD, Principal Investigator — Saiseikai Yokohama City Eastern Hospital
Locations (2):
- Japan (2):
  - Edogawa Hospital, Tokyo
  - Saiseikai Yokohama City Eastern Hospital, Yokohama